CLINICAL TRIAL: NCT06602661
Title: A Prospective Randomized Study of Reinforced Vs Non-reinforced Staple Lines in Fissureless Lobectomy
Brief Title: Reinforced and Non-Reinforced Staple Lines in Fissureless Lobectomy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Surrey Thoracic Surgery Group (Other)
Collaborators: Johnson and Johnson Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6997
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Lung; Lung Adenocarcinoma; Lung Adenosquamous Carcinoma; Lung Cancer, Non-Small Cell; Lung Carcinoma; Lobectomy; Lobectomy Patient; Lobectomy by Video-thoracoscopies; VATS
Keywords: Prospective Randomized Study; Fissureless Lobectomy; Prolonged Air Leak (PAL); Pulmonary Resections; Hospital Length of Stay (LOS); Lung Carcinoma; Echelon 3000 stapler; Endopath Stapler Line Reinforcement; Video-Assisted Thoracoscopic Surgery (VATS); Postoperative Outcomes; Intraoperative Characteristics; Randomized Control Trial (RCT); Surrey Memorial Hospital (SMH); Surrey Thoracic Surgery Group (STSG); Digital Drainage System (Thopaz); Chest Tube Duration; Hospital Readmission; Patient Outcomes; Bioabsorbable Buttress Material; Polyglactin and Polydioxanone
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fissureless Lobectomy with Non-Reinforced Staple Lines Using ECHELON™ 3000 (Active Comparator): Arm Description: Participants in the control arm will undergo fissureless lobectomy using the ECHELON™ 3000 stapler without any reinforcement. This intervention involves: Thorough patient assessment and confirmation of eligibility criteria. Informed consent process emphasizing the use of non-reinforced staplers. Standard general anesthesia with double lumen endotracheal tube and patient positioning for lobectomy. Utilization of video-assisted thoracoscopic surgery (VATS). Division of pulmonary artery branches, veins, and bronchus with non-reinforced stapler. Division of lung parenchyma using the ECHELON™ 3000 stapler without reinforcement. Placement of chest tube size 28 Fr for all patients. Standard postoperative monitoring in the recovery room and monitored bed afterward. Implementation of standardized pain management protocols. Regular assessment for air leaks and drainage amount using a digital drainage system (Thopaz). Performing daily chest X-rays (CXR) until tube removal.
  Interventions: Procedure: Fissureless Lobectomy with Non-Reinforced Staple Lines
- Fissureless Lobectomy with Reinforced Staple Lines Using ECHELON™ 3000 and ENDOPATH™ Reinforcement (Experimental): Participants in the experimental arm will undergo fissureless lobectomy using the ECHELON™ 3000 stapler equipped with the ENDOPATH™ stapler line reinforcement. This intervention involves:Thorough patient assessment and confirmation of eligibility criteria. Informed consent process emphasizing the use of reinforced staplers. Standard general anesthesia with double lumen endotracheal tube and patient positioning for lobectomy. Utilization of video-assisted thoracoscopic surgery (VATS). Division of pulmonary artery branches, veins, and bronchus with non-reinforced stapler. Division of lung parenchyma using the ECHELON™ 3000 stapler with ENDOPATH™ reinforcement. Placement of chest tube size 28 Fr for all patients. Standard postoperative monitoring in the recovery room and monitored bed afterward. Implementation of standardized pain management protocols. Assessment for air leaks and drainage amount using a digital drainage system (Thopaz). Performing daily chest X-rays (CXR) until removal.
  Interventions: Procedure: Fissureless Lobectomy with Reinforced Staple Lines

INTERVENTIONS:
Procedure: Fissureless Lobectomy with Reinforced Staple Lines — This intervention involves performing a fissureless lobectomy, a type of lung surgery where the lobes of the lung are removed without dissecting the fissures between them. The procedure utilizes the ECHELON™ 3000 stapler equipped with the ENDOPATH™ stapler line reinforcement. The ENDOPATH™ device uses bioabsorbable buttress material made from Polyglactin and Polydioxanone, designed to enhance the durability and effectiveness of the staple line.
  The reinforcement tool is a novel preloaded device with a "click and go" mechanism, making it easy to load and use during surgery.
  The primary objective is to reduce the average duration of hospital length of stay (LOS) directly caused by prolonged air leak (PAL). Secondary objectives include improving intraoperative characteristics (such as duration and amount of blood loss) and postoperative outcomes (such as incidence and duration of PALs, number of chest tube days, and incidence of hospital.
  Arms: Fissureless Lobectomy with Reinforced Staple Lines Using ECHELON™ 3000 and ENDOPATH™ Reinforcement
Procedure: Fissureless Lobectomy with Non-Reinforced Staple Lines — This intervention involves performing a fissureless lobectomy, a type of lung surgery where the lobes of the lung are removed without dissecting the fissures between them. The procedure utilizes the ECHELON™ 3000 stapler without any additional reinforcement. This means the staple lines are created using the standard stapler without the use of bioabsorbable buttress materials.
  The ECHELON™ 3000 stapler is used to divide the lung parenchyma, pulmonary artery branches, veins, and bronchus without any reinforcement, relying solely on the standard stapling mechanism.
  Arms: Fissureless Lobectomy with Non-Reinforced Staple Lines Using ECHELON™ 3000

SUMMARY:
Prolonged Air Leak (PAL) is a common and serious problem after lung surgery. It can lead to worse patient outcomes, longer hospital stays, and higher costs. Reinforced staplers are designed to make the staple line stronger and reduce the risk of PAL. However, investigators don't know if they are better than standard staplers, especially in a specific type of lung surgery called fissureless lobectomy for lung cancer. This study aims to find out if reinforced staplers are more effective at reducing PAL and its complications compared to non-reinforced staplers.

Reinforced staplers have been used in lung surgeries and have shown to reduce PAL. For example, staplers with special materials like polyglycolic acid (PGA) sheets have shown lower air leakage and fewer days with chest tubes. Other materials like expanded polytetrafluoroethylene (ePTFE) sleeves have also been used to manage air leaks in different types of lung surgeries. However, their effectiveness in fissureless lobectomy has not been studied yet.

DETAILED DESCRIPTION:
The standard definition of a PAL by the Society of Thoracic Surgeons (STS) dictates that the leak persists beyond five days; however, clinical practices commonly broaden this definition to include any instances in which the leak delays hospital discharge. Some studies find that air leaks persisting after 72 hours are indicative of PAL. Therefore, investigators have elected to use 72 hours as our benchmark for this study.

In addition to an increased hospital LOS, PAL can heighten costs, increase the incidence of readmission, and induce other postoperative complications. PAL is therefore one of the most significant complications for patients undergoing pulmonary resections, particularly lobectomy for lung cancer. PAL remains a problem despite enhancements in endoscopic surgical techniques; consequently, reinforced staplers have been developed to provide additional support to the staple line, thereby enhancing its sealing capabilities.

Reinforced staplers have been used in pulmonary surgeries, including lobectomies, and the results have shown a reduction in PAL occurrence. For example, staplers with polyglycolic acid (PGA) sheets demonstrated a lower postoperative air leakage rate and a reduction in number of chest tube days. Another study reported application of expanded polytetrafluoroethylene (ePTFE) sleeves in the management of air leaks following thoracoscopic and open lung volume reduction surgery.

The comparative effectiveness of reinforced versus non-reinforced staplers in the context of fissureless lobectomy has not yet been established. By implementing a randomized control trial design, this prospective study will attempt to fill this knowledge gap and uncover the ability of reinforced staplers to improve patient outcomes. To quantify these effects, hospital LOS will be used as a primary measure. Additional intraoperative and postoperative characteristics will be used to document any secondary benefits to reinforced staplers regarding their safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over.
* Patients undergoing fissureless lobectomy for lung carcinoma.

Exclusion Criteria:

* Patients suitable for sub lobar resections.
* Patients undergoing lobectomy for indications other than lung cancer.
* Patients with a history of pleural adhesions.
* Patients with previous lung resection on the same side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Length of Stay Due to Prolonged Air Leak (PAL) | Up to 30 days post- surgery
  1. The primary objective is to determine whether the use of reinforced staple lines in fissureless lobectomies will reduce the average duration of hospital length of stay directly caused by prolonged air leaks.
  -measured in days

SECONDARY OUTCOMES:
Intraoperative Characteristics and Postoperative Outcomes | Within 30 days post-surgery
  1. The number or percentage of patients experiencing prolonged air leaks postoperatively.
  * measured by number or Percentage 2. The duration of prolonged air leaks in days.
  * Measured in Days 3. The total number of days each patient has a chest tube in place postoperatively.
  * Measured in Days 4. The number or percentage of patients readmitted to the hospital within 30 days post-surgery.
  * Measured in number or Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Surrey Thoracic Surgery Group, Surrey, B.C, Canada

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD: This encompasses all data gathered during the study, including preoperative, intraoperative, and postoperative variables.
  IPD that underlie results in a publication: This includes data that directly support the findings and conclusions presented in any resulting publications from the study.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD and supporting information will be available starting from January 1, 2028.
Access Criteria: * Qualified researchers affiliated with academic, medical, or research institutions.
  * Healthcare professionals involved in related clinical research or patient care.
  * Regulatory authorities for the purpose of regulatory review and compliance.
  They Will Be Able to Access:
  * De-identified Individual Participant Data (IPD), including demographic information, clinical outcomes, and other relevant variables.
  * Supporting information such as study protocols, statistical analysis plans, and informed consent forms.
  How They Will Be Able to Access It:
  * Interested parties must submit a formal request to the Principal Investigator (PI) at Dr. Ahmad S. Ashrafi.
  * Upon approval, a data use agreement (DUA) must be signed.
  * Approved researchers will access the data through a secure, password-protected online platform.

REFERENCES:
- See also: Early Postoperative Complications — https://ebook.sts.org/sts/view/Pearsons-General-Thoracic/1418125/all/Early_Postoperative_Complications
- See also: Endobronchial Valves in Treatment of Persistent Air Leak — https://pubmed.ncbi.nlm.nih.gov/38870914/
- See also: Estimating hospital costs attributable to prolonged air leak in pulmonary lobectomy — https://pubmed.ncbi.nlm.nih.gov/15691691/
- See also: A Novel, Easy-to-Use Staple Line Reinforcement for Surgical Staplers — https://pubmed.ncbi.nlm.nih.gov/32099487/
- Available data/document: Study Protocol — https://docs.google.com/document/d/1-NMx1lP-_x1KHA0t49yEG7tNsFgepmyWPkbdFfWMPMc/edit?usp=sharing
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1rON8VADRvws1J_I_rmqAAy2sNgL0I9c5/view?usp=sharing